CLINICAL TRIAL: NCT00666094
Title: A Randomized Controlled Trial of Strength Versus Aerobic Exercise Training to Improve Glycemic Control in Men With Type 2-diabetes
Brief Title: A Randomized Controlled Trial of Exercise Training Among Men With Type 2-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 520073168; 520073168 (Other: SVT)
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia
Keywords: Type 2-diabetes; exercise therapy; RCT; Norway
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Endurance Training; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endurance training (Active Comparator): supervised endurance training
  Interventions: Behavioral: Endurance training
- strength training (Experimental): Supervised strength training
  Interventions: Behavioral: strength training

INTERVENTIONS:
Behavioral: Endurance training — supervised endurance training. Three sessions per week in three months.
  Other Names: Aerobic training
  Arms: endurance training
Behavioral: strength training — Supervised strength training. Three sessions per week in three months.
  Arms: strength training

SUMMARY:
To test the hypothesis that there is no difference in change in HbA1C among men with type 2-diabetes after an exercise intervention with strength versus endurance training.

DETAILED DESCRIPTION:
Exercise training is well documented as part of effective treatment for type 2-diabetes patients. Endurance training has been suggested as the most suitable form of exercise. There are reasons to believe that strength training also has a positive effect. However, comparisons of endurance training and strength training regimes are limited.

Therefore we randomized 26 men with type 2-diabetes to either an endurance training group or a strength training group. Both groups exercised three sessions per week for three months. The training was supervised.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2-diabetes
* Male, 35-71 years
* Managing their diabetes through a lifestyle and/or the drug metformin only
* Able to participate in either of the exercise groups

Exclusion Criteria:

* Symptomatic cardiovascular disease
* Uncontrolled hypertension
* Physical or cognitive disabilities that will interfere with participating in the exercise regimes.
* Trained consistently during the last six months.

Ages: 35 Years to 71 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
HbA1C | 12.01.08

SECONDARY OUTCOMES:
body composition, C-peptid, BP, Cholesterol (LDL, HDL), Triglycerides | 12.01.08

CONTACTS AND LOCATIONS:
Overall Officials: Liv B Augestad, PhD, Study Director — National Taiwan Normal University
Locations (1):
- NTNU, Trondheim, Norway

REFERENCES:
- [Result] Moe B, Augestad LB, Åsvold BO, Flanders WD. Effects of aerobic versus resistance training on glycaemic control in men with type 2 diabetes. European Journal of Sports Science 11(5): 365-374, 2011